CLINICAL TRIAL: NCT05495737
Title: A Pragmatic Randomized Control Trial of Nurse-Delivered Brief Meaning Centered Psychotherapy for Homebound Palliative Care Patients
Brief Title: Meaning-Centered Psychotherapy at Home
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 22-019
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Nurse-Patient Relations; Psychology, Social
Keywords: Meaning Centered Psychotherapy; Meaning Centered Psychotherapy for Palliative Patients; 22-019; Memorial Sloan Kettering Cancer Center
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Phase 1: Nurse Participants: n=8-10 nurses
  Interventions: Behavioral: Meaning-Centered Psychotherapy/MCP-PC Training
- Phase 1: Patient Participants: n=8-10 patients
  Interventions: Behavioral: Meaning-Centered Psychotherapy/MCP-PC
- Phase 2: Nurse Participants: n=8-10 nurses
  Interventions: Behavioral: Meaning-Centered Psychotherapy/MCP-PC Training
- Phase 2: Patient Participants Meaning-Centered Psychotherapy/MCP-PC Intervention Arm: n=35
  Interventions: Behavioral: Meaning-Centered Psychotherapy/MCP-PC
- Phase 2: Patient Participants Treatment As Usual/TAU Intervention Arm: n=35
  Interventions: Behavioral: Treatment As Usual/TAU

INTERVENTIONS:
Behavioral: Meaning-Centered Psychotherapy/MCP-PC Training — Two-Day MCP-PC Training for Nurses (including mock patient/simulation with actor) with a Pre- and Post-Training Assessment
  Groups: Phase 1: Nurse Participants; Phase 2: Nurse Participants
Behavioral: Meaning-Centered Psychotherapy/MCP-PC — 3 sessions, completed over the course of 3-6 weeks in the participant's home
  Groups: Phase 1: Patient Participants; Phase 2: Patient Participants Meaning-Centered Psychotherapy/MCP-PC Intervention Arm
Behavioral: Treatment As Usual/TAU — Research team will provide:
  1. feedback about level of distress at time of screening
  2. local referral for psychological care
  Groups: Phase 2: Patient Participants Treatment As Usual/TAU Intervention Arm

SUMMARY:
The purpose of this study is to train nurses from the VNS Health Visiting Nurse Service to deliver Meaning-Centered Psychotherapy for Palliative Care Patients (MCP-PC) to homebound people, and to evaluate how effective MCP-PC is for people with cancer.

ELIGIBILITY:
Participant Inclusion Criteria:

Nurses (all phases):

* Per self-report, providing direct care services at VNS Health
* Per self-report, fluent in English**
* Per self-report, is age 18 or older

Patients (all phases):

* Per health record and/or self-report, is a patient in the VNS Health home health agency division (post-acute care)
* Per health record and/or self-report, is age 18 or older
* Per health record, has a cancer diagnosis and a rating of ≥ 2 on Symptom Control Scale
* Per health record and/or self-report, fluent in English**
* Has a score of ≥ 4 on Callahan cognitive screener
* Has a score of ≥ 4 on Distress Thermometer (N/A for Training Case Participants)

  * Language verification: For both nurses and patients, prior to enrollment, all will be asked the following two questions by a Clinical Research Coordinator (CRC) to verify

English fluency necessary for participation in the study:

1. How well do you speak English? (must respond "very well" or "well" when given the choices of Very well, Well, Not well, Not at all, Don't know, or Refused)
2. What is your preferred language for healthcare? (must respond English)

Participant Exclusion Criteria:

Nurses (all phases):

* Per self-report, planning to leave position at VNS Health in the next 6 months

Patients (all phases):

* Per health record and/or self-report, has a diagnosis of Alzheimer's, dementia, or other organic brain disorder and in the judgment of the PIs is unable to meaningfully participate.
* Per health record, has impaired decision-making capacity
* Per health record and/or self-report, is permanently placed in a nursing home
* Per health record and/or self-report, is currently receiving Hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both patients and homecare nurses will be recruited and enrolled as participants in the proposed study. All participants will be recruited from VNS Health Visiting Nurse Service
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2026-08-08 (Estimated); Study Completion 2026-08-08 (Estimated)

PRIMARY OUTCOMES:
MPI Competency Ratings | 2 years
  Phase I portion: To refine the MCP-PC training and study procedures for homecare delivery by nurse interventionists as determined by providers' MPI Competency Ratings

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Saracina, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Visiting Nurse Service of NY, New York, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Saracino RM, Park EY, Onorato N, Pessin H, McDonald M, Demirjian C, Schofield E, Rosenfeld B, Breitbart W, Applebaum AJ. A pragmatic randomized controlled trial of nurse-delivered brief Meaning Centered Psychotherapy at Home (MCP-H) for individuals with advanced cancer: Study protocol. J Geriatr Oncol. 2025 Nov;16(8):102736. doi: 10.1016/j.jgo.2025.102736. Epub 2025 Oct 3. PMID 41045824
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

DOCUMENTS (1):
  • Informed Consent Form (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT05495737/ICF_000.pdf